CLINICAL TRIAL: NCT05661760
Title: Development of a Clinical Prediction Model to Facilitate Decision Making in Interdisciplinary Biopsychosocial Rehabilitation in Patients With Osteoarthritis (OA)
Brief Title: Predicting Successful Outcome of Interdisciplinary Biopsychosocial Rehabilitation in Osteoarthritis
Acronym: CIR-predict
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University (Other)
Collaborators: Centrum voor Integrale Revalidatie (CIR) (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CIR-001; 41150323011N (Other: CAPHRI-Maastricht University)
Record Dates: First submitted 2022-11-24; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Chronic Pain; Osteoarthritis; Disability Physical
Keywords: multimodal treatment; interdisciplinary; rehabilitation medicine; prediction model; treatment outcome
MeSH Terms: conditions — Chronic Pain; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic pain osteoarthritis: Patients with chronic pain and disability with osteoarthritis
  Interventions: Behavioral: interdisciplinary multimodal pain treatment

INTERVENTIONS:
Behavioral: interdisciplinary multimodal pain treatment — A combination of physical and psychosocial treatment methods is employed, including Emotional Awareness and Expression Therapy (EAET), Pain Neuroscience Education (PNE), Acceptance and Commitment Therapy (ACT), graded activity, exposure in vivo, and experiential learning through physical training.
  Other Names: biopsychosocial treatment

SUMMARY:
The goal of this prospective study is to identify variables that can predict whether an interdisciplinary biopsychosocial intervention for patients with osteoarthritis will be successful.

Using an observational design, patients admitted to this program during the 3-year period (2019-2021) will be included and data gathered during routine clinical practice at baseline and end of treatment of patients who gave informed consent, will be used.

With these data a prediction model will be build and internal validation with bootstrapping will be done.

DETAILED DESCRIPTION:
Rationale: To predict the probability of a positive outcome of interdisciplinary biopsychosocial intervention in individual patients with osteoarthritis (OA), a prediction model is needed.

Research Question/Objective: The overall goal is to develop a clinical prediction model to facilitate decision making in interdisciplinary biopsychosocial rehabilitation in patients with OA. The model will predict the individual probability (in percentage) of a positive response to the treatment (treatment success).

Design: A retrospective cohort design. Setting: A Dutch rehabilitation facility. Participants: Patients with OA diagnosed by a medical specialist and consisting at least three months.

Intervention and procedures: The intervention of interest is interdisciplinary biopsychosocial rehabilitation. The procedures include the development of a clinical prediction model and assessment of its performance and internal validity.

Measurements: Candidate predictors will be carefully selected. The outcome of the model will be treatment success, defined by the change on the Pain Disability Index (PDI). The model will be built with data gathered as part of routine practice.

Expected outcome of the research: The deliverable will be a clinical predication model, which can be used in follow-up research.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain > 3 months and osteoarthritis
* Large personal and social dysfunction
* Interplay of biological, social and psychological factors maintaining pain and/or disability

Exclusion criteria:

* Inability to actively participate in treatment (insufficient motivation, limited Dutch language skills, environmental factors, other pending treatments)
* Disagreement between patient and care providers on content of treatment
* Pending legal procedures that hinder full cooperation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Referred by GP, medical specialist or occupation physician to reduce level of disability and improve quality of life of patients fulfilling the eligibility criteria and not having one or more of the exclusion criteria:
Sampling Method: Probability Sample
Enrollment: 2309 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Disability Index | baseline (start of treatment) and 10 weeks
  Measures to which degree pain prevents the patient from participating in daily activities. Improvement equal or higher than Minimal Clinically Important Change (MCID; which is 9 points) is defined as successful treatment, and all others as not successful treatment Population will be dichotomized into successful or non-successful treatment and this will be the dependent variable for the logistic regression analysis used to build the prediction model

OTHER OUTCOMES:
Brief Illness Perception Questionnaire | Baseline
  Measures the cognitive and emotional representation of illness in a patient
Pain Self Efficacy Questionnaire | baseline
  Measures how confident the patient is that he/she will be able to perform daily tasks despite being in pain
Psychological Inflexibility in Pain Scale | Baseline
  Measures psychological inflexibility (avoidance of pain and cognitive fusion with pain)
Symptom Checklist 90 | Baseline
  Measures to which degree the patient suffers from 90 different physical and psychological symptoms.
Hospital Anxiety and Depression Scale | Baseline
  Measures feelings of fear and depression, without looking at physical complaints
General CIR questionnaire | baseline
  Records general socio-demographic characteristics as well as symptom-related information, co-morbidity and medication levels.
Pain Catastrophising Scale | Baseline
  Measures degree of catastrophizing
Checklist Individual Strength | Baseline
  Measures subjective tiredness
Twelve-Item Short Form Health Survey | Baseline
  Measures physical and mental functioning
Patient Specific Complaint | Baseline
  Measures a patient's functional status by inquiring for three self-selected daily activities to which degree the patient is limited in this activity by his/her pain complaints

CONTACTS AND LOCATIONS:
Overall Officials: Rob J Smeets, MD PhD, Principal Investigator — Maastricht University
Locations (1):
- Centrum voor Integrale Revalidatie, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
As data are gathered as routine practice, data are owned by and stored by CIR. In case of any request the PI can be contacted and he will ask CIR whether specific data will be made available

REFERENCES:
- [Background] Breugelmans L, Scheffer E, Beckers LWME, Oosterwijk RFA, Nijland G, Smeets RJEM. Systematic description of an interdisciplinary multimodal pain treatment programme for patients with chronic musculoskeletal pain, using the TIDieR checklist. BMC Res Notes. 2022 Oct 11;15(1):320. doi: 10.1186/s13104-022-06211-z. PMID 36221116